CLINICAL TRIAL: NCT03497858
Title: The Effect of Coconut Water on Varsity Basketball Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Dr. Peter Lemon, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111166
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Water; Gatorade; Coconut Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- coconut water (Experimental): participants will complete the simulated basketball game with coconut water supplementation
  Interventions: Other: Coconut Water
- Placebo - water (Placebo Comparator): participants will complete the simulated basketball game with water supplementation
  Interventions: Other: Placebo - water
- Sports drink (Experimental): participants will complete the simulated basketball game with sports drink supplementation
  Interventions: Other: Sports drink

INTERVENTIONS:
Other: Coconut Water — participants will consume coconut water and complete a simulated basketball game
  Arms: coconut water
Other: Placebo - water — participants will consume Placebo - water and complete a simulated basketball game
  Arms: Placebo - water
Other: Sports drink — participants will consume a sports drink and complete a simulated basketball game
  Arms: Sports drink

SUMMARY:
This study will assess whether there is a performance enhancing effect associated with hydrating with coconut water. There have been only two studies in the past that have examined this phenomenon, however these studies have limitations due to their design parameters. Kalman et al. (2012) ".... while treadmill time to exhaustion is routinely used in laboratory studies, the use of a time trial test as the measure of exercise performance may be more appropriate." While Peart et al. (2016) stated: "limitations to the exercise protocol employed here may have contributed to the absence of a performance improvement with coconut water."

DETAILED DESCRIPTION:
Purpose The purpose of the study is to determine whether hydrating with coconut water during a game-simulated, basketball-specific training session can enhance performance. It is hypothesized that coconut water will provide an ergogenic effect for basketball players.

Sample The sample will include 20 varsity basketball players, male and female, ranging in age from 18-35 who volunteer to participate in the study. This sample size is justified assuming a standard deviation of 1.5 based on previous studies and using a power of 80% with the statistical significance of 0.05 the resulting n would be 2(1.5)^2*(0.84+1.96)^2/5=7 (Kadam, P., & Bhalerao, S. (2010). Sample size calculation. International journal of Ayurveda research, 1(1), 55). To account for dropouts, 10 participants will be recruited for each group. Participants will be required to have no history of kidney problems. All individuals must give written informed consent in order to participate in the study. Exclusion criteria include not being a varsity basketball player, being younger than 18 or older than 35, or having a history of kidney problems.

Procedure Inclusion/exclusion criteria will be explicitly stated throughout the recruitment process. Potential participants will be recruited through first contacting the Men's and Women's Head Basketball Coaches of Western University and obtaining approval of collaboration from the team. Players will then be in direct contact with Reed Zehr to gain information of study. After given the study details, individuals will be given up to 3 days to determine if they want to participate and give their informed consent. See attached form in the consent section of the ethics application.

Measurement: All players will perform two sessions of a 10 minute BSST (Basketball Specific Skills Test) which will represent the 1st and 2nd quarter respectively. Field Goal Attempts (FGA) (#), Field Goals Made (FGM) (#), Field Goal Percentage (FGP) (%) will be measured from the free-throw line, mid-range and three point distances during the BSST. A dribbling drill will be used as well and number of dribbles (#) will be measured. All players will then perform two sessions of a 10 minute BEST (Basketball Exercise Simulation Test) test which will represent the 3rd and 4th quarter of a basketball game. Total distance covered (m), Mean circuit completion time (s), mean sprint time (s), and total sprint decrement (%) will be measured during the BEST.

Protocol: On test days, participants will report to he Gym at 0600 h after a 12 h overnight fast and having abstained from any strenuous exercise following the evening meal. At 0615 h, participants will consume a standardized breakfast (toast and jam) and the first beverage of 750mL. At 0730 h, participants will be told to consume the second beverage of 250mL. At 0745 h, the participants will undergo the first 10 min quarter of the BSST. At 0755 h, the participants rest during a 2 min break (1st intermission) and consume the third beverage of 250mL. At 0757 h, the participants will undergo the second session of the BSST. At 0807 h, the participants receive a 15 min break (half-time) and consume the fourth beverage of 500mL. At 0822 h, the participants will undergo the first BEST. At 0832 h, the participants receive a 2 min break (2nd intermission) and consume the final beverage of 250mL. At 0834 h, the participants undergo the second BEST. At 0844, the exercise bout will be completed. Participants will complete this protocol for each of the three experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-35 years old
* Must be a Canadian Varsity Basketball Player

Exclusion Criteria:

* Younger than 18 or older than 35
* Not a Canadian Varsity Basketball Player

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Field Goal Percentage | 16 mins
  shots made / shots attempted X 100
Dribbles Performed | 5 minutes
  number bounces
Total Sprint Decrement | 20 mins
  100 x (total sprint time / ideal sprint time) - 100
Distance run | 20 mins
  meteres run

SECONDARY OUTCOMES:
Rating of Perceived Exertion | 2 mins
  Subjective rating from 6-20, 6 being easy and 20 being very, very hard

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Exercise Nutrition Laboratory (Western University), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kalman DS, Feldman S, Krieger DR, Bloomer RJ. Comparison of coconut water and a carbohydrate-electrolyte sport drink on measures of hydration and physical performance in exercise-trained men. J Int Soc Sports Nutr. 2012 Jan 18;9(1):1. doi: 10.1186/1550-2783-9-1. PMID 22257640